CLINICAL TRIAL: NCT03064672
Title: Transcervical Balloon Catheters in GBS Carriers, Is It Safe? A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BALLOONGBS- HMO-CTIL
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-08

CONDITIONS: GBS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- induction by transcervical Balloon Catheters insertion (Experimental)
  Interventions: Device: transcervical Balloon Catheters
- induction without transcervical Balloon Catheters (No Intervention)

INTERVENTIONS:
Device: transcervical Balloon Catheters — induction of labor by transcervical Balloon Catheters insertion
  Arms: induction by transcervical Balloon Catheters insertion

SUMMARY:
This prospective cohort study aims to determine whether maternal and neonatal outcomes are affected by GBS carrier status in women undergoing transcervical balloon catheter insertion.

ELIGIBILITY:
Inclusion Criteria:

* During the study period and in the absence of contraindications, women anticipating induction of labor with unripe cervix will be screened for eligibility.
* Inclusion criteria are singleton gestation with confirmed cephalic presentation
* Gestational age between 37+0/7 and 41+6/7 weeks'
* Intact membranes
* Reactive non-stress test and Bishop's score < 6.

Exclusion Criteria:

* Women less than 18 years, with multiple gestation pregnancies, pregnancies with major fetal anomalies, vaginal infection, intrauterine fetal death and those who were not candidates for vaginal delivery (placenta previa, non-cephalic presentation, planned cesarean delivery).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
adverse neonatal outcomes | 2-3 days
  the incidence of composite adverse neonatal outcomes based on the NICE criteria for early detection of neonatal sepsis

SECONDARY OUTCOMES:
composite adverse maternal outcomes | 2-3 days
  chorioamnionitis, suspected chorioamnionitis or endometritis, urinary tract infection or sepsis in the peripartum period, prolonged hospital stay, and allergic reaction to antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Doron Kabiri, MD, Study Director — Hadassah Medical Organization

IPD SHARING:
Plan to Share IPD: No
The data of the mother and the baby will be checked and recorded. At the end of the study, all the data are gonna be analyzed. In case of a severe bad outcome, the data will be checked during the study to make sure that the study is not the cause.

REFERENCES:
- [Background] Kabiri D, Hants Y, Yarkoni TR, Shaulof E, Friedman SE, Paltiel O, Nir-Paz R, Aljamal WE, Ezra Y. Antepartum Membrane Stripping in GBS Carriers, Is It Safe? (The STRIP-G Study). PLoS One. 2015 Dec 31;10(12):e0145905. doi: 10.1371/journal.pone.0145905. eCollection 2015. PMID 26719985